CLINICAL TRIAL: NCT04994275
Title: Impact of Iron Deficiency on the Incidence of Postoperative Infections - CARIPO Observational Study
Brief Title: Impact of Iron Deficiency on the Incidence of Postoperative Infections
Acronym: CARIPO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202100105
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Iron-deficiency; Postoperative Complications; Postoperative Infection
Keywords: iron-deficiency; infection; postoperative; major surgery
MeSH Terms: conditions — Anemia, Iron-Deficiency; Postoperative Complications; Infections | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to undergo a major elective surgery
  Interventions: Other: no intervention, but presence of ID or not

INTERVENTIONS:
Other: no intervention, but presence of ID or not — This is an observational study regarding patients admitted to undergo a major elective surgery supposed to last more than an hour. Investigators will analyzed the incidence of postoperative infections up to 90 days after surgery according to the preoperative iron status: iron deficiency (defined as a ferritin of less than 100 µg/L or <300 µg/L And TSAT<20%) or no iron deficiency

SUMMARY:
Iron deficiency is a common state during the perioperative period. Data from literature do not allow us to conclude on how perioperative iron deficiency influences postoperative infections occurrence. This prospective observational study aims to assessed the postoperative infections incidence according to the preoperative iron-stock status.

DETAILED DESCRIPTION:
Postoperative infections are one of the most common complication after surgery, involving 2 to 50% of patients according to series and representing 16% of healthcare associated infections. Postoperative infections are highly morbid and result in a significant cost for the society, by increasing the length of hospital stay for example. They also have an impact on bacterial ecology because of the use of broad-spectrum antibiotic therapy to treat nosocomial infection. The decrease of postoperative infections occurrence is a major public health challenge.

Iron deficiency, with or without iron-deficiency anemia, is also very common during the perioperative period. Its prevalence goes from 30 to 40% and even up to 60% when associated with anemia. Iron deficiency is associated with an increased morbidity and mortality. Indeed, iron is a mineral element essential for oxygen transport through hemoglobin, but also implied in cellular metabolism by its role in the electron transport chain and in the citric acid cycle in the mitochondrion. Hence, iron is essential for the proper functioning of the immune system. Iron deficiency leads to an alteration of cellular immune defenses with a decrease in neutrophils function secondary to reduced myeloperoxidase activity, an alteration of their phagocytic capacity, a decrease in the number of T lymphocytes and a weaker response to antigenic exposure, an alteration of Natural Killer lymphocytes activity and a lower interleukine-2 production by lymphocytes. Thus, iron deficiency was associated with an increased risk of sepsis in human.

According to an old cohort published in 1988, a preoperative iron deficiency (defined by ferritin ≤20 ng/L) on 448 patients who underwent abdominal surgery, was associated with an increased in postoperative infections (23 vs 5 infections, p<0,001) and with a longer hospital stay (12±4 vs 8±3 days, p<0,001). However, a recent prospective observational study (2018), regarding orthopedic elective surgery, iron deficiency was not associated with an increased perioperative morbidity nor mortality. The statistical power was limited (100 patients, whose 6 only with iron deficiency, postoperative infections are rare in elective orthopedic surgery and assessed at day 30 instead of day 90 as recommended).

Accordingly, data from literature do not allow us to conclude on how perioperative iron deficiency influences postoperative infections occurrence. Yet, patients might benefit from preoperative iron supplementation. The PREVENTT randomized controlled trial, published in October 2020, studied the impact of intravenous iron supplementation before major abdominal surgery for anemic patients. This trial found a statistically significant decrease in hospital readmission in the treatment group and a downward trend in the occurrence of postoperative infections. Similar results were highlighted in 2016 in a randomized controlled trial comparing the fate of patients according to iron supplementation or not immediately after surgery.

Those results invite to undertake further clinical studies to better characterize the impact of iron deficiency and its correction on postoperative infections occurrence.

Our first hypothesis is that preoperative iron deficiency would be associated with an increased incidence of postoperative infections after major surgery and that its correction would lessen this association.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Iron-deficiency assessment realized by blood sample as part of standard care
* Elective surgery supposed to last more than an hour

Exclusion Criteria:

* Adult under tutelage
* Emergency surgery
* Refusal of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult admitted to undergo elective surgery supposed to last more than an hour and who had an iron-deficiency assessment realized by blood sample as part of standard care
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative infectious complication | 90 days
  The main goal of this study is to compare the incidence of postoperative infectious complications according to the preoperative patient's iron-stock status (supplemented or not). The primary outcome is the occurrence of at least one infection complication within 90 days after surgery.
  The various infections recorded are defined by the Center for disease control and prevention and included:
  * superficial surgical site infection (within 30 days after surgery) or deep surgical site infection (within 30 days after surgery or 90 days if an implant is in place)
  * pneumonia
  * urinary infection
  * bacteriemia
  * catheter infection

SECONDARY OUTCOMES:
To assess the prevalence of preoperative iron deficiency according to the surgical field | Preoperative
To assess the incidence of postoperative infections according to the type of surgery | 90 days
  The various infections recorded are defined by the Center for disease control and prevention and included:
  * superficial surgical site infection (within 30 days after surgery) or deep surgical site infection (within 30 days after surgery or 90 days if an implant is in place)
  * pneumonia
  * urinary infection
  * bacteriemia
  * catheter infection
To assess the incidence of overall postoperative complications according to the iron-stock status | 90 days
  Postoperative complications are assessed by the POMS (Postoperative Morbidity Survey)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France